CLINICAL TRIAL: NCT01480791
Title: A Double-Blind, Randomized, Parallel Design Study of Aliskiren Versus Hydrochlorothiazide in Mild-to Moderate Hypertensive Type II Diabetes Mellitus Patients on Remodeling of Resistance Arteries
Brief Title: Aliskiren vs Hydrochlorothiazide in Hypertensive Type II Diabetic Patients on Resistance Arteries
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Because of results of Altitude trial, this trial was cancelled.
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Ernesto L. Schiffrin, Physician-in-Chief, Director of the Cardiovascular Prevention Center, Professor of Medicine, McGill University, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSPP100ACA03T
Record Dates: First submitted 2011-11-05; First posted 2011-11-29 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Hypertension; Diabetes
Keywords: resistance arteries; endothelial dysfunction; aortic stiffness
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — aliskiren; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hydrochlorothiazide (Active Comparator): Treatment of patients with hydrochlorothiazide and effect on small arteries
  Interventions: Drug: Hydrochlorothiazide
- Aliskiren (Experimental): Treatment of patients with aliskiren and effect on small arteries
  Interventions: Drug: Aliskiren vs. hydrochlorothiazide; Drug: Hydrochlorothiazide
- Normotensive non diabetic subjects (No Intervention): A comparator non intervention normotensive non diabetic group of healthy subjects will be used for baseline comparison of primary and secondary endpoints

INTERVENTIONS:
Drug: Aliskiren vs. hydrochlorothiazide — Aliskiren will be used at increasing doses from 150 to 300 mg per day for 6-12 months.
  Other Names: Aliskiren is Tekturna or Rasilez
  Arms: Aliskiren
Drug: Hydrochlorothiazide — Hydrochlorothiazide will be used at increasing doses from 12.5 to 25 mg per day for 6-12 months.
  Other Names: Hydrochlorothiazide is a generic drug.
  Arms: Aliskiren; Hydrochlorothiazide

SUMMARY:
This study will be performed only at the Jewish General Hospital. It will investigate the effect of treatment with aliskiren, an inhibitor of renin, a substance produced by the kidney that constricts arteries and raises blood pressure, on the blood vessels, specifically the arteries, of subjects who have diabetes and elevated blood pressure (hypertension).

To investigate blood vessels, different techniques will be used. For large arteries, these will be studied by non invasive methods using detection of the pulse wave or using ultrasound over the skin of the neck, the wrist and the groin. To study small vessels, the investigators will perform a biopsy on the buttock, under local anesthesia, and obtain a small sample of tissue from under the skin, from which the vessels will be dissected. The investigators have performed many hundreds of these small biopsies over the past 20 years for similar studies without any complications. The biopsies are very well tolerated. From this research the investigators will thus be able to learn what the structure and function of these vessels is in these patients, in comparison to a normal healthy group.

The hypertensive diabetic subjects will then be assigned by chance (randomized trial) to treatment with the renin inhibitor aliskiren or a comparator, the diuretic hydrochlorothiazide. Aliskiren is a relatively new drug used to treat hypertension that is very well tolerated and is now being evaluated in numerous trials in hypertensive diabetic individuals. The diuretic is a well-know agent used to treat high blood pressure now for many years, and which is very well tolerated. Physicians, nurses and scientists involved in the study will be unaware of who is receiving which drug, as will be the patients (this is the meaning of double-blind trial). However, if there is any problem, the secret code will be broken and the individual withdrawn from the study. Subjects will be treated for a year, and the study procedures (non invasive and the biopsy) repeated at 6 months and after one year of treatment. During the study, blood samples will be drawn and urine collected at certain intervals to ensure safety of the treatment.

Once tissues are obtained they will be studied in the laboratory. The study of the vessels will allow treatment us to determine how the treatment with the renin inhibitor aliskiren affects the structure and function as well as cellular and molecular aspects of arteries of hypertensive diabetic persons. The investigators expect these studies to provide us knowledge on mechanisms and perhaps new targets for future therapies of cardiovascular disease and hypertension.

ELIGIBILITY:
Inclusion Criteria:

Hypertensive Group

* Diabetes mellitus (diagnosed for at least 6 months) will be defined by usual criteria based on basal glycemia or glucose tolerance test . Diabetes must be well controlled, with glycosylated hemoglobin below 0.08 (8%).
* Hypertension is defined as a mean SiSBP > 130 mmHg or SiDBP of 85-115mmHg at the screening visit, and after two weeks of placebo therapy. (Hypertension will be considered essential if there is no evidence of an underlying treatable cause after suitable clinical and laboratory assessment. Hypertensive patients may be taking any antihypertensive agent except a renin inhibitor. They may be taking an ACE inhibitor or an ARB, which will not be discontinued. If they have been on HCTZ, they are eligible to participate.
* Subjects are 30-70 years old
* Informed Consent obtained by patient

Criteria for inclusion: Control Group

* Diabetic defined as: hemoglobin A1C < 0.06 ( 6%) and / or fasting glycemia < 5.6mmol/L.
* Hypertensive defined as : SiSBP ≤120 mmHg and/or SiDBP ≤80mmHg
* Subjects are 30-70 years old
* Informed Consent obtained by patient

Exclusion Criteria:

* Uncontrolled diabetes ( defined as: preprandial glycemia usually above 10 mmol/L and glycosylated hemoglobin above 0.08).
* Renovascular hypertension
* History of malignant hypertension
* Sitting systolic blood pressure > 210 mmHg
* Cerebrovascular accident within the past year, or current transient ischemic attacks
* History of myocardial infarction, percutaneous coronary angioplasty or coronary artery bypass surgery
* Clinically significant AV conduction disturbances and/or arrhythmias (e.g. second- or third-degree AV block; Sick-sinus syndrome or clinically significant bradycardia- resting heart rate < 45 beats/minute).
* Tachyarrhythmias; clinically significant arrhythmias
* Presence of an accessory bypass tract (e.g. Wolff-Parkinson-White syndrome)
* Angina pectoris
* Current or prior history of heart failure or known left ventricular ejection fraction ≤ 40%
* History of unexplained syncope or a known syncopal disorder (e.g., Stokes-Adams Syndrome)
* Presence or known history of hemodynamically significant obstructive valvular disease or hypertrophic cardiomyopathy
* Hypertensive patients already taking a renin inhibitor.

Concomitant treatment

* Psychotropic or Antidepressant Agents
* Major psychotropic agents such as phenothiazines are not permitted. Chronic doses of antidepressants are not permitted.
* Oral Contraceptives are not allowed if the patient's hypertension was induced by this medication.
* Regular use of NSAID is permitted if taken regularly on a stable regimen. Aspirin in small doses (≤ 1 g/day) as a cardioprotective agent is permitted. Acetaminophen is permitted.
* Other Drugs
* Concomitant use of oral or inhaled steroids, ACTH, immunosuppressants or lithium are not allowed, nor are cyclosporine, quinidine, aliskiren available from the market.

Laboratory Parameters

* Glycosylated hemoglobin above 0.08 (8%).
* Plasma creatinine concentration ≥ 200 μmol/L (adjusted for age and weight).
* Prior to patient entry, any hematuria should be evaluated, the etiology established/documented, and treatment rendered as appropriate.
* Off-treatment serum potassium concentration ≥ 5.5 mmol/L or ≤ 3.5 mmol/L
* AST (SGOT) or ALT (SGPT) > 2 x normal upper limit, and if clinically significant
* Clinically significant laboratory values outside of the established normal range including but not limited to any of the following parameters: hematocrit, hemoglobin, platelet count or white blood cell count
* Allergies/Hypersensitivity /Pulmonary
* Known hypersensitivity or contraindication to aliskiren or thiazide diuretics.
* History of clinically important malabsorption or gastrointestinal resection.
* Smoking of 10 cigarettes or more is excluded. Also excluded are co-existent conditions which could independently affect the histology of resistance vessels except for diabetes (e.g. any disease which may be associated with vasculitides: collagen-vascular diseases, chronic hepatitis B antigenemia, circulating immune complexes, complement disorders, amyloidosis, scleroderma, etc.).
* Pregnancy or lactating females. Females of childbearing age who are not surgically sterilized and who are using effective contraception may enter only if an exclusionary pregnancy test is done within 72 hours of the first double-blind dose of test agent. Pregnancy tests will then be done monthly throughout the study in women capable of conception.
* Other concurrent severe disease which could preclude participation or survival, such as neoplasm or Acquired Immunodeficiency Syndrome (AIDS), or patients known to be HIV positive.
* Any known bleeding or platelet disorder.
* The known absence of one kidney.
* Patients who are currently abusing or previously abused alcohol or other drug substances (within past two years).
* Mentally or legally incapacitated patients.
* Patients who have participated in another investigational drug trial, including those using marketed drugs (i.e. patient has signed a consent form), within the 28 days prior to start of placebo therapy.
* Patients who, in the opinion of the investigator, will not cooperate fully, keep appointments or are generally unreliable.
* Inability or unwillingness on the part of the patient to sign the Patient Consent Form.
* Phase V of Korotkoff sounds cannot be detected.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is baseline-adjusted change in media/lumen ratio in patients who were randomized to aliskiren (group 1) comparatively to those randomized to hydrochlorothiazide (group 2) | 6 months-1 year
  The primary endpoint is baseline-adjusted change in media/lumen ratio in patients who were randomized to aliskiren (group 1) comparatively to those randomized to hydrochlorothiazide (group 2)

SECONDARY OUTCOMES:
Secondary outcome: Pulse wave velocity (PWV) of aorta in hypertensive diabetic patients randomized to aliskiren versus those who were randomized to HCTZ. | 6 months-1 year
  Pulse wave velocity (PWV) of aorta in hypertensive diabetic patients randomized to aliskiren versus those who were randomized to HCTZ.
Augmentation index (AI) of patients randomized to either aliskiren or hydrochlorothiazide | 6 months-1 year
  Evaluation by non invasive means with a SphygmoCor of augmentation index (AI) of central aortic blood pressure in response to either aliskiren or hydrochlorothiazide in hypertensive diabetic patients.
Flow-mediated dilation in hypertensive diabetic patients randomized to aliskiren vs. hydrochlorothiazide | 6 months-1 year
  Evaluation by non invasive means with ultrasound of flow-mediated dilation of the brachial artery in response to either aliskiren or hydrochlorothiazide in hypertensive diabetic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto L Schiffrin, MD, PhD, Principal Investigator — SMBD-Jewish General Hospital
Locations (1):
- Cardiovascular Prevention Centre, Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Schiffrin EL, Park JB, Intengan HD, Touyz RM. Correction of arterial structure and endothelial dysfunction in human essential hypertension by the angiotensin receptor antagonist losartan. Circulation. 2000 Apr 11;101(14):1653-9. doi: 10.1161/01.cir.101.14.1653. PMID 10758046
- [Background] Savoia C, Touyz RM, Endemann DH, Pu Q, Ko EA, De Ciuceis C, Schiffrin EL. Angiotensin receptor blocker added to previous antihypertensive agents on arteries of diabetic hypertensive patients. Hypertension. 2006 Aug;48(2):271-7. doi: 10.1161/01.HYP.0000230234.84356.36. Epub 2006 Jun 19. PMID 16785331
- [Background] Savoia C, Touyz RM, Amiri F, Schiffrin EL. Selective mineralocorticoid receptor blocker eplerenone reduces resistance artery stiffness in hypertensive patients. Hypertension. 2008 Feb;51(2):432-9. doi: 10.1161/HYPERTENSIONAHA.107.103267. Epub 2008 Jan 14. PMID 18195160
- See also: Web page of Dr. Ernesto L. Schiffrin at Lady Davis Institute for Medical Research — http://www.ladydavis.ca/en/ernestoschiffrin